CLINICAL TRIAL: NCT00446693
Title: A Single Arm, Multi-center, Prospective Clinical Investigation to Evaluate Safety and Performance of the EndoFast Reliant™ System in Vaginal Wall Reinforcement
Brief Title: Clinical Investigation to Evaluate Safety and Performance of the EndoFast Reliant™ System in Vaginal Wall Reinforcement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endogun Medical Systems Ltd. (Industry)
Responsible Party: Dr. Miron Livneh VP Clinical and Medical affairs, Endogun Medical Systems Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFPS01
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Use of EndoFast Reliant System
  Interventions: Device: EndoFast Reliant™ system for Pelvic Organ Prolapse repair

INTERVENTIONS:
Device: EndoFast Reliant™ system for Pelvic Organ Prolapse repair — The EndoFast Reliant™ system is a new concept of reinforcing the vaginal wall with proprietary mesh and soft-tissue Fasteners in a minimally-invasive procedure.

SUMMARY:
The purpose of this study is to clinically assess the safety and performance of the EndoFast Reliant™ system as a less invasive treatment for Pelvic Organ Prolapse.

DETAILED DESCRIPTION:
Background:

Pelvic Organ Prolapse represents a significant problem worldwide and may have a significant negative impact on a woman's quality of life. The uterus, rectum and the bladder are held in their normal positions just above the inner end of the vagina by a "hammock" made up of supportive muscles and ligaments. Wear and tear on these supportive structures in the pelvis can allow the uterus, the bladder, the bowels, the vaginal vault or the rectum to sag through the muscle and ligament layers. When this occurs, the rectum, uterus, bowels or bladder can create a bulge into the vagina. In severe cases, it is possible for the sagging rectum, uterus, bowels or bladder to work its way down far enough that the bulge can appear at the vagina's opening or even protrude from the opening. Pelvic Organ Prolapse causes significant discomfort to the patients being associated with urinary incontinence, voiding difficulty culminating with urinary retention, constipation, pain during sexual intercourse, local discomfort, etc.

Treatment Options When symptoms occur, many patients initially opt for conservative treatment. Pelvic exercises and vaginal support are the current mainstays of non surgical management. In addition, patients who are poor surgical candidates or are strongly disinclined to surgery can be offered vaginal support (pessaries) for symptom relief. Topical estrogen is an important adjunct in the conservative management of patients with Pelvic Organ Prolapse. However, the primary management strategy for severe Pelvic Organ Prolapse is surgical. The exact treatment choice will depend on the severity of the prolapse and whether there are any related pelvic floor defects.

Endogun Medical Systems Ltd. has developed an innovative, minimally-invasive system for repair of Pelvic Floor Prolapse. The EndoFast Reliant™ system is a new concept of reinforcing the vaginal wall with a proprietary system comprised of a mesh and soft tissue fasteners in a minimally-invasive way. The fasteners can be deployed easily and swiftly in narrow spaces into soft tissue and can support substantially more weight than needed for Pelvic Organ Prolapse repair. Following many pre-clinical tests, the EndoFast Reliant™ system is now available for clinical evaluation.

The objective of this study is to evaluate the safety and performance of the EndoFast Reliant™ system for treatment of Pelvic Organ Prolapse.

In particular:

* The study's primary goal is to clinically assess the safety of the EndoFast Reliant™ as a minimally-invasive procedure for vaginal wall reinforcement.
* The study's secondary goal is to clinically evaluate the performance of the EndoFast Reliant™ system as a minimally-invasive procedure for vaginal wall reinforcement by evaluating the improvement in Pelvic Organ Prolapse using the POPQ grading system.

Study Procedures and Follow up:

Pre-treatment tests and inspection will be performed within 4 months prior to surgery.

Approximately two weeks, three months and six months after the surgery the patient will be invited for physician examination and laboratory tests.

Additional Study Measures:

In addition to the endpoint parameters, the following study measures will be collected:

* Symptoms relief and Quality of Life (QOL) considerations.
* Sexual Function considerations, as documented using the Female Sexual Function (FSFI) questionnaire;
* Assessment of the physician's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 40-80 years (inclusive) who is not pregnant or planning to have further births.
* Subject suffers from Pelvic Organ Prolapse confirmed by vaginal inspection.
* Patient under reliable form of contraceptive measure or menopausal.
* Subject able to comprehend procedure and has signed Informed Consent Form for participation in this study.
* Subject able to complete the applicable questionnaires.

Exclusion Criteria:

* Planned to undergo hysterectomy.
* Uterine prolapse equal to or greater than 3rd degree.
* Documented Stress Urinary Incontinence on physical examination with full bladder or during complete urodynamic assessment with and without prolapse reduction.
* Any chronic active and uncontrolled disease.
* Vaginal bleeding disorders.
* Needing emergency surgery.
* Any acute disease.
* Blood clotting disorders and/or anticoagulant treatment.
* Known cognitive or psychiatric disorder.
* High operative risk.
* Any ongoing malignant disease.
* Concurrent participation in any other clinical trial

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety is defined as paucity of major device-related complications. | 12 months

SECONDARY OUTCOMES:
Performance as defined by relative improvement in Pelvic Organ Prolapse staging (as reported post operatively versus preoperatively) using the POPQ grading system. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Von Theobald, Prof., Principal Investigator — Professeur d'Université-Praticien Hospitalier, gynécologie; Michel Cosson, Prof., Principal Investigator — Hôpital Jeanne de Flandre - CHRU Gynécologie obstétrique; Genadi Bitman, MD, Principal Investigator — Sheba Medical Center
Locations (3):
- France (2):
  - CHU de Caen, Caen
  - Hôpital Jeanne de Flandre - CHRU Gynécologie obstétrique, Lille
- Sheba Medical Center, Ramat Gan, Israel